CLINICAL TRIAL: NCT03751774
Title: The National Danish MAMAACT Intervention
Brief Title: The MAMAACT Intervention
Acronym: MAMAACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: 19 maternity wards (Ambiguous); Migrant medical clinics (Odense and Hvidovre) (Unknown); TrygFonden, Denmark (Industry); Østifterne (Unknown); Danske Regioner (Other); Neighbourhood mothers (Unknown); University College Copenhagen (Other)
Responsible Party: Principal Investigator, Sarah Fredsted Villadsen, Assistant Professor / Ph.D, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAMAACT
Record Dates: First submitted 2018-11-12; First posted 2018-11-23 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Health Literacy; Stillbirth; Apgar; 0-3 at 1 Minute; Apgar; 4-7 at 1 Minute; Asphyxia
MeSH Terms: conditions — Stillbirth; Asphyxia

STUDY DESIGN:
Intervention Model Description: Clusters (maternity wards) are randomized to either intervention or control (standard ANC). Intervention coverage 27000. Data collection for the primary and secondary trial outcomes includes 1.921 interviewed participants in the pre-intervention survey and 2.232 interviewed participants in the post-intervention survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAMAACT (Experimental): Training of midwives in intercultural communication. A 6 hours course and 2 one hour booster sessions. Distribution of health education materials on warnings signs of pregnancy and health system navigation to pregnant women during antenatal care visits.
  Interventions: Behavioral: MAMAACT
- Control (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: MAMAACT — Post graduate training and health education materials
  Arms: MAMAACT

SUMMARY:
Inequalities in stillbirth, infant and child mortality as well as other reproductive health outcomes have been reported among ethnic minority groups in Denmark. The MAMAACT study aims to improve the communication between non-Western immigrant women and midwives regarding body symptoms that need prompt reaction, and thus improve perinatal health. 19 of 21 maternity wards in Denmark participate in the study. By simple randomization 10 maternity wards have been selected to the intervention group and 9 maternity wards to the control group. The intervention consist of post graduate training of midwives in intercultural competence and use of health education materials (leaflet and app) on pregnancy warning signs. The intervention will be implemented in the antenatal care from October 2018- September 2019. The training is expected to reach 350 midwives working with antenatal care and 27000 pregnant women, of whom 2700 are expected to be non-Western migrant women. The effect of the MAMAACT intervention will be analyzed by assessing women's ability to actively engage with health care providers (primary outcome), women's knowledge about warning signs of pregnancy complications and health system navigation using survey data. Secondary outcomes are 5-minute Apgar score, umbilical-cord blood gas analysis, transfer to a neonatal intensive care unit, gestational age at birth, fetal birthweight according to gestational age and ICD-10 code for sign of asphyxia.

MAMAACTs overall target group is all pregnant women, and the specific target group is women of non-Western origin. Therefore, the outcomes of the trial will be analysed for both the total population and for the effects among non-Western immigrant women specifically.

Hypothesis: Training of midwives in intercultural competence and increased attention to communication of warning signs of pregnancy during antenatal care will improve the communication and interaction between women and midwives, improve health literacy of the women and enable them to better access the relevant care in case of a pregnancy complication, which will then increase survival and health of newborn children.

DETAILED DESCRIPTION:
The intervention is a complex intervention and designed as a cluster randomised trial. 19 maternity wards participate and by simple randomization within thee groups of maternity wards according to the proportion of non-Western migrant women giving birth, 10 clusters are in the intervention group and 9 in the control group.

The effectiveness of the intervention will be analysed in a difference-in-difference design, where the change in outcomes from before to after intervention period at the intervention sites are compared to the change at the control sites. Cross sectional surveys will be conducted before and after the implementation of the intervention.

Participants for the pre-implementation survey will be enrolled from May to July 2018. Participants for the post-implementation survey will be enrolled from May to July 2019. Only participants from the post-implementation survey at the intervention sites will be exposed to the intervention. The start date for the enrollment of participants exposed to the intervention will therefore be May 1st 2019.

The primary trial outcome is studied using telephone surveys with pregnant women recruited through the antenatal care services. The questionnaire will include validated items on the health literacy dimension actively engagement with health care providers (5 items) and health system navigation (5 items). Women are recruited when they attend for the week 20 ultra sound scan and will be interviewed between pregnancy week 30+0 and 38+7. The questionnaires are managed in six languages (Danish, Arabic, English, Turkish, Somali and Urdu, and bilingual and trained interviewers conduct the interviews.

Using unpublished data from pregnant women at Hvidovre Hospital in 2016 (n=407), Danish born women are found to have a mean level of the relevant health literacy dimension on 4.16 and non-Western migrant women have a significantly lower mean at 3.97. The goal is that the MAMAACT intervention will to improve the mean level of the non-Western migrant women to the level of the Danish born women at baseline, thus an effect on 0.2 on the mean of the dimension are to be shown. A recent Danish cluster randomized trial aiming at improved breast feeding by improving the guidance of new mothers at maternity wards has reported intra-cluster correlation coefficients (ICC) under 0.005.

For the sample size calculation an estimation with 10 cluster in the control group and 10 clusters in the intervention group were used, however after recruitment and randomization 9 wards were in the control group and 10 in the intervention group. With an ICC on 0.005 with 10 clusters in the intervention arm and 10 clusters in the control arm an effect on 0.1 with a strength of 80 % can be detected if data from 2580 of the total population before and after the intervention (1290 from the intervention before and after and 1290 from the control group before and after) is collected.

With an ICC on 0.005 with 10 clusters in the intervention arm and 10 clusters in the control arm an effect on 0.2 with a strength of 80 % can be detected if data is collected from 500 non-Western women before and after the intervention (250 from the intervention both before and after and 250 from the control group both before and after).

Based on telephone survey data, effects on the skills in health system navigation among the women will also be analysed.

The overall effects of the MAMAACT intervention on stillbirth and neonatal health will be analysed by the medical birth registry and obstetric databases. Stillbirth is defined as death of a child without any signs of life after 22 completed weeks of gestation. Neonatal death is defined as death of a child after live birth before 1 months of age. No significant effects on these outcomes are expected due to low numbers in the short intervention period. Secondary trial outcomes are 5-minute Apgar score, umbilical-cord blood gas analysis, transfer to a neonatal intensive care unit, gestational age at birth, fetal birthweight according to gestational age, ICD-10 code for sign of asphyxia, and pregnancy complications (preeclampsia).

All effectiveness analysis will be using an intention-to-treat approach and will account for the clustering of individuals and potential confounding in a controlled mixed effect regression.

The implementation of the intervention will be analyzed using qualitative data. The resarch questions are: How do midwives and non-Western immigrant women react to the MAMAACT intervention across Denmark? Which barriers exist in the organisation of antenatal care, and how do they affect the national implementation of the MAMAACT intervention? What are non-Western immigrant women's everyday life conditions in Denmark, and how do they affect women's responses to potential pregnancy complications?

ELIGIBILITY:
Inclusion Criteria:

* Clusters: All maternity wards in Denmark defined as having one midwife heading the unit. Thus, Odense and Svendborg maternity wards are considered one cluster
* Survey: Women attending the malformation scan in the specified calender weeks at the specific maternity ward, pregnancy week 18+0 to 22+0 during the malformation scan, able to participate in a phone interview in Danish, Arabic, English, Turkish, Somali or Urdu

Exclusion Criteria:

* Cluster: All maternity wards invited
* Survey: Women out of the gestational age range specified above, women who could not speak the selected languages

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Enrollment: 4153 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Actively engagement with health care providers | Assessed among women in prenancy week 30+0 to 38+7
  Increased mean score of the domain (5 item scale) among non-Western migrant women in Denmark. The Health Literacy domain of Actively engagement with health care providers, validated in the Health Literacy Questionnaire

SECONDARY OUTCOMES:
Apgar score at 5 minutes | Mean Apgar scores at five minutes after birth
  Increased mean of apgar score at 5 minutes among non-Western migrant women. Using nation wide registers
Ability to navigate the health system | Assessed among women in pregnancy week 30+0 to 38+7
  Increased ability to navigate the health system among non-Western migrant, women assessed using the validated Health Literacy Questionnaire domain on Health System Navigation (5 item scale)
Knowledge on pregnancy warning signs | Assessed among women in pregnancy week 30+0 to 38+7
  Increased knowledge on what to do in case of vaginal bleeding, severe headache and deep vein thrombosis during pregnancy among non-Western migrant women. Survey data
Umbilical-cord blood gas analysis | Umbilical-cord blood gas analysis taken after the delivery of the baby, within the 30 minutes
  Improvements in the mean umbilical-cord blood gas levels as signs of asphyxia for non-Western migrant women in a time phase before the intervention with the period of implementation. Using nation wide registers
Transfer to a neonatal intensive care unit | Transferral at the day of delivery or the day after
  Reduced number of non-Western new born children admitted to neonatal unit. Using nation wide registers
ICD-10 code for sign of asphyxia | Assessed within the first minute after delivery
  Reduced number of non-Western children having the ICD10 code for sign of asphyxia. Using nation wide registers
Maternal pregnancy complications | Assessed from pregnancy week 12 up till one week after delivery
  Reduced proportion of severe maternal pregnancy complications, focus on preeclampsia
A composite score for stillbirth, neonatal death and neonatal near miss | Assessed according to the specific outcomes with the maximum range of 28 days after birth for neonatal death
  The composite score is defined as having one or more of the following outcomes: stillbirth, neonatal death (death at age 0-28 completed days from birth) and the infant focused outcomes above (outcome 2 (apgar score at 5 minutes), 5 (umbilical-cord blood gas ), 6 (transfer to a neonatal intensive care unit) and 7(ICD-10 code for sign of asphyxia)).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah F Villadsen, Ph.d., Principal Investigator — University of Copenhagen
Locations (19):
- Denmark (19):
  - The maternity ward in Aabenraa, Sygehus Soenderjylland, Aabenraa
  - The maternity ward in Aalborg, Aalborg Universitetshospital, Aalborg
  - The maternity ward in Aarhus, Aarhus Universitetshospital, Aarhus
  - The maternity ward in Esbjerg, Sydvestjysk Sygehus, Esbjerg
  - The maternity ward in Herlev, Herlev Hospital, Herlev
  - The maternity ward in Herning, Hospitalsenheden Vest, Herning
  - The maternity ward in Hillerød, Nordsjællandshospital Hillerød, Hillerød
  - The maternity ward in Hjoerring, Regionshospitalet Nord, Hjørring
  - The maternity ward in Holbaek, Holbaek Sygehus, Holbæk
  - The maternity ward in Horsens, Regionshospitalet Horsens, Horsens
  - The maternity ward in Hvidovre, Hvidovre hospital, Hvidovre
  - The maternity ward in Kolding, Sygehus Lillebaelt, Kolding
  - The maternity ward in Nykøbing Falster, Nykøbing Falster Sygehus, Nykøbing Falster
  - The maternity ward in Næstved, Næstved Sygehus, Næstved
  - The maternity ward in Odense, Odense Universitetshospital, Odense
  - The maternity ward in Randers, Regionshospitalet Randers, Randers
  - The maternity ward in Roskilde, Sjaellands Universitetshospital Roskilde, Roskilde
  - The maternity ward in Bornholm, Bornholms Hospital, Rønne
  - The maternity ward in Viborg, Regionshospitalet Viborg, Viborg

REFERENCES:
- [Derived] Rasmussen TD, Nybo Andersen AM, Ekstrom CT, Jervelund SS, Villadsen SF. Improving health literacy responsiveness to reduce ethnic and social disparity in stillbirth and infant health: A cluster randomized controlled effectiveness trial of the MAMAACT intervention. Int J Nurs Stud. 2023 Aug;144:104505. doi: 10.1016/j.ijnurstu.2023.104505. Epub 2023 May 1. PMID 37267853